CLINICAL TRIAL: NCT06875557
Title: MIND MATTERS; UNVEILING THE IMPACT OF DIGITAL MENTAL HEALTH INTERVENTION (DMHI) ON PSYCHOLOGICAL DISTRESS AMONG YOUTH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Madeeha Fatima, Principal Investigator, Fatima Jinnah Women University
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FJWU/EC/2024/92
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-04

CONDITIONS: Psychological Distress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional : who receives intervention i.e., Digital Mental Health Intervention (DMHI) (Experimental): Digital Mental Health Intervention (DMHI) was provided to the sample of young adults who were experiencing psychological distress. DMHI was being given through Insight Timer application that only focused on reiki healing techniques. Insight Timer is a mobile app that provides guided meditations to calm the mind, alleviate anxiety, manage stress, achieve deep sleep, and enhance well-being and happiness. Additionally, it offers calm and soothing music, educational courses, live events, and workshops in multiple languages. (Insight Network, Inc., n.d.). The app is FREE to download with an email allowing access to their collection of meditation recordings. Insight Timer's free-to-use feature is most suitable for community groups.
  Interventions: Behavioral: Digital Mental Health Intervention (DMHI)
- Waitlist Control : who would receive intervention after the study completion (Active Comparator): Digital Mental Health Intervention (DMHI) was provided to the sample of young adults who were experiencing psychological distress. DMHI was being given through Insight Timer application that only focused on reiki healing techniques. Insight Timer is a mobile app that provides guided meditations to calm the mind, alleviate anxiety, manage stress, achieve deep sleep, and enhance well-being and happiness. Additionally, it offers calm and soothing music, educational courses, live events, and workshops in multiple languages. (Insight Network, Inc., n.d.). The app is FREE to download with an email allowing access to their collection of meditation recordings. Insight Timer's free-to-use feature is most suitable for community groups.
  Interventions: Behavioral: Digital Mental Health Intervention (DMHI)

INTERVENTIONS:
Behavioral: Digital Mental Health Intervention (DMHI) — In the current study, the impact of Digital Mental Health Intervention (DMHI) would be examined through Insight Timer application, focusing on just its one aspect (Reiki healing techniques). Through the usage of DMHIs in the young population, youth would be better able to express their psychological issues with the healthcare professionals instead of the fear of being labelled or stigmatization.
  Arms: Interventional : who receives intervention i.e., Digital Mental Health Intervention (DMHI)
Behavioral: Digital Mental Health Intervention (DMHI) — Digital Mental Health Intervention (DMHI) was provided to the sample of young adults who were experiencing psychological distress. DMHI was being given through Insight Timer application that only focused on reiki healing techniques. Insight Timer is a mobile app that provides guided meditations to calm the mind, alleviate anxiety, manage stress, achieve deep sleep, and enhance well-being and happiness. Additionally, it offers calm and soothing music, educational courses, live events, and workshops in multiple languages. (Insight Network, Inc., n.d.). The app is FREE to download with an email allowing access to their collection of meditation recordings. Insight Timer's free-to-use feature is most suitable for community groups.
  Arms: Waitlist Control : who would receive intervention after the study completion

SUMMARY:
The current study would be designed to identify the impact of digital mental health intervention on psychological distress among youth through Insight Timer app focusing on reiki healing techniques. Furthermore, in this study, the predictors such as Childhood Trauma, Type-D personality and Substance Abuse would be studied that will be associated with psychological distress among youth. Moreover, the study will also focus on the mediating role of Type-D personality in the relationship between childhood trauma and psychological distress, and substance abuse and psychological distress, as indicated by existing theories and literature (Luo et al., 2022; Javakhishvili & Widom, 2021). The study will further investigate the effectiveness of Digital Mental Health Intervention (DMHI) for type-D personality and childhood trauma (emotional abuse, physical abuse, sexual abuse, emotional neglect, physical neglect).

DETAILED DESCRIPTION:
The current study will be designed to assess the efficacy of digital mental health intervention for the management of psychological distress among youth in Pakistan. The study will also examine the mediating role of Type-D personality in the relationship between childhood trauma/ substance abuse and psychological distress. The study will be conducted in two phases. Phase 1 will be a cross-sectional survey and phase 2 will be a randomized controlled trial. A sample of 367 young adults (aged 15-24 years) would be recruited for the cross-sectional survey from different institutions of Rawalpindi and Islamabad. In the 2nd phase, selected young adults will be equally divided into interventional (25 participants) and control group (25 participants). Type-D personality, childhood trauma, substance abuse and psychological distress will be measured with DS-14, CTQ-28, DAST-10, DASS-21 respectively. Type-D personality, childhood trauma, substance abuse will be identified as significant predictors of psychological distress. In phase 2 (RCT), the intervention group will receive an 8-week Digital Mental Health Intervention (DMHI), whereas the control group will not receive any intervention. This research will contribute to the growing literature on the benefits of digital mental health apps, suggesting DMHIs as a viable non-pharmacological approach in alleviating psychological distress among youth. It would underscore the importance of integrating digital mental health apps in mental health interventions, especially in cultures and contexts like Pakistan, where such approaches are emerging. .

ELIGIBILITY:
Inclusion Criteria: Young boys and girls ranging from 15 to 24 years and those who agreed to participate in the study, not have been diagnosed with any chronic physical or mental illness were included as sample for the study, particularly all those respondents who were fluent in English language (as mode of language used in the questionnaires and the Digital Mental Health Intervention) and own an iPhone, iPad, iPod or smartphone with access to the internet.

- Exclusion Criteria: Participants excluded from the study were those who did not fulfil the inclusion criteria: Young boys and girls under the age of 15 years and above 24 years as well as those who didn't had access to smartphone, iPad, iPhone or any other such device; unavailability of internet service; those who were suffering from any severe psychiatric illness, either in the present or in the past; especially those who were on medication or treatment for such problem in the last one year; those suffering from any deliberating physical disease or disability, either in the present or in the past; those who were on any kind of long-term medication for any disease or disorder; as these all can negatively affect the results of the study.

-

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 376 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale (DASS-21) | 2 months
  Depression Anxiety and Scale Scale (DASS-21, Lovibond & Lovibond, 1995; was used to assess psychological distress in terms of depression, anxiety and stress in the participants. It contains 21 items with three 7-items subscales; depression (item number 3, 5, 10, 13, 16, 17 and 21), anxiety (item number 2, 4, 7, 9, 15, 19 and 20) and stress (1, 6, 8, 11, 12, 14 and 18). Participants responded on a Likert scale which ranged from 0 i.e., "did not apply to me at all" to selecting 3 i.e., "applied to me very much, or most of the time". It assessed the degree to which symptoms had been present in the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Madeeha Fatima Fatima, M.Phil Scholar, Principal Investigator — Fatima Jinnah Women University
Locations (1):
- Fatima Jinnah Women University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to some ethical concerns, the gathered data will not be shared. All research findings will be published in an anonymous way in an aggregated form.

REFERENCES:
- See also: Denollet, J. (2005). DS14: Standard assessment of negative affectivity, social inhibition, and Type D personality. Psychosomatic Medicine, 67(1), 89-97. https://doi.org/10.1097/01.psy.0000149256.81953.49 — https://doi.org/10.1097/01.psy.0000149256.81953.49